CLINICAL TRIAL: NCT05324618
Title: A Comparative Clinical Trial to Evaluate the Efficacy and Safety of Tacrolimus Versus Hydrocortisone in Treatment of Children With Atopic Dermatitis
Brief Title: Tacrolimus Versus Hydrocortisone in Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: National Hepatology & Tropical Medicine Research Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Tacrolimus vs Hydrocortisone
Record Dates: First submitted 2022-01-16; First posted 2022-04-12 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2022-01

CONDITIONS: Atopic; Dermatitis
Keywords: Tacrolimus; Hydrocortisone; Atopic; Dermatits; children
MeSH Terms: conditions — Dermatitis | interventions — Tacrolimus; Pharmaceutical Preparations; Chemical Industry; Hydrocortisone

STUDY DESIGN:
Intervention Model Description: prospective, double blinded, simply randomized clinical trial
Who Masked: Participant, Care Provider
Masking Description: 200 opaque envelopes will be numbered serially and the corresponding letter which denotes the allocation will be put according to the electronic randomization table. Then all envelopes will be closed and put in one box. When the first patient arrives, the envelope will be opened and the patient will be allocated according to the letter inside.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tacrolimus group (Active Comparator): 100 patients treated by thin layer of 0.03% topical tacrolimus ointment on the affected areas twice daily for 4 months.
  Interventions: Drug: Tacrolimus
- Hydrocortisone group (Active Comparator): 100 patients treated by thin layer of 1% hydrocortisone cream on the affected areas twice daily for 4 months.
  Interventions: Drug: Hydrocortisone

INTERVENTIONS:
Drug: Tacrolimus — 0.03% topical tacrolimus ointment applied on the affected areas twice daily for 4 months.
  Other Names: Tacrolimus (Tacrolimus 0.03%®) was manufactured by AL-Andalous company for pharmaceutical and chemical industries, Egypt.
  Arms: Tacrolimus group
Drug: Hydrocortisone — 1% hydrocortisone cream applied on the affected areas twice daily for 4 months.
  Other Names: Hydrocortisone (Micort 1%®) was manufactured by Cid company for pharmaceutical and chemical industries, Egypt.
  Arms: Hydrocortisone group

SUMMARY:
Atopic dermatitis (AD) is a very common inflammatory, genetic skin disorder that occurs more frequently in children. Its exact etiology is not known but it is characterized by pruritic skin reactions with elevation in the levels of inflammatory markers. Corticosteroids are the first line and the mainstay therapy in management of atopic dermatitis but have many local and systemic adverse effects. The study aims to evaluate the efficacy and safety of topical tacrolimus ointment in comparison to topical hydrocortisone cream in management of children diagnosed with atopic dermatitis.

DETAILED DESCRIPTION:
Atopic dermatitis is a common pruritic inflammatory skin disorder. The prevalence of atopic dermatitis increased in the last three decades by two or three folds worldwide. In the developed countries, atopic dermatitis is estimated to affect 15% to 30% of children and 2% to 10% of adults. This type of dermatitis is usually associated with family history of other atopic disorders such as allergic rhinitis or asthma.

The clinical presentation of Atopic dermatitis differs depending on the age of the patient, it usually begins in infancy with erythematous, papular skin rash that may first appear on the cheeks and chin. In childhood, the skin appears dry, flaky, rough, cracked, and may bleed because of scratching, in adults the lesions are more diffuse with underlying erythema.

This condition is characterized by acute phase where the skin has red scaly patches and chronic phase in which the skin thickens.

Atopic dermatitis is a complex genetic disease where the exact etiology is not entirely known, but it is most probably due to interaction between environmental and genetic factors. The two major groups of involved genes are the genes encoding for epidermal and epithelial structural proteins and the genes regulating the production of cytokines for the immune response.

In atopic dermatitis patients, imbalance occurs between T helper-1 (TH1) and T helper-2 (TH2) immune responses, increased TH2 activity causes the release of interleukin (IL)-3, IL-4, IL-5, IL-10, and IL-13 which results in blood eosinophilia, increased total serum immunoglobulin (Ig) E, and increased growth and development of mast cells.

Atopic dermatitis patients are more likely to develop different skin infections as compared to healthy individuals, including: staphylococcal secondary bacterial infections and herpes simplex viral infection.

Topical corticosteroids (TCS) are the mainstay for management of atopic dermatitis to which other treatments are compared, they act by many pathways to reduce inflammation. Although TCS are effective treatment, they have both local adverse effects as skin thinning, striae, perioral dermatitis, acne, rosacea, telangiectasias, purpura and focal hypertrichosis. Moreover, systemic absorption can lead to systemic effects such as hypothalamic-pituitary-adrenal (HPA) axis suppression, infections, hyperglycemia, cataracts, glaucoma, and growth retardation (in children).

All these side effects are more likely to occur with prolonged use and so seeking for other treatment options is crucial.

Topical calcineurin inhibitors (TCI) as tacrolimus and pimecrolimus are immunosuppressives that help to control the acute flares and decrease the severity of the new flares by acting as immunomodulators. They inhibit the calcineurin so inhibit the T-cell proliferation that produces many inflammatory cytokines such as IL-2, IL-3, IL-4, IL-17, tumor necrosis factor (TNF). TCI is more selective as compared to TCS with less adverse effects so it is considered as an acceptable alternative to TCS.

Tacrolimus 0.03% ointment is approved for moderate to severe atopic dermatitis for ages 2 years and older, with the 0.1% ointment limited to ages 16 years and older; pimecrolimus 1% cream is approved for mild-to-moderate atopic dermatitis for ages 2 years and older. There is limited data comparing TCS with tacrolimus or pimecrolimus.

The FDA has a black box warning for both tacrolimus ointment and pimecrolimus cream about their potential local skin carcinogenesis as seen in animal studies. However, till now there is no causal relationship has been proven between use of a TCI and the development of lymphoma or non-melanoma skin cancer.

This study aims to assess the efficacy and safety of topical tacrolimus ointment in comparison to topical hydrocortisone cream in children diagnosed with atopic dermatitis. The primary outcome is to evaluate the effect of topical tacrolimus ointment as compared to topical hydrocortisone cream by estimation of the serum level of inflammatory cytokines and the effect on the dermatitis severity scale. The secondary outcome is to evaluate the tacrolimus safety as compared to hydrocortisone through the assessment of treatment related toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients
* 2-16 years old
* diagnosed with Atopic Dermatitis according to Hanifin and Rajka criteria

Exclusion Criteria:

* patients with serious skin disorder other than Atopic Dermatitis
* patients taking systemic corticosteroids or anti-inflammatory medications.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
evaluate the effect of topical tacrolimus ointment as compared to topical hydrocortisone cream on the serum level of different inflammatory cytokines using enzyme linked immunosorbent assay technique (ELISA) | 4 months
  estimation of the serum level of inflammatory cytokines (biochemical evaluation of IL-10 (pg/ml), IL-17 (pg/ml), IL-23 (pg/ml) using enzyme linked immunosorbent assay technique (ELISA)
severity assessment | 4 months
  Estimation of the effect on the dermatitis severity scale using the modified Eczema Area and Severity Index (mEASI) score. It is a tool used to evaluate the severity of eczema based on body surface area affected by lesions, morphology of lesions (erythema, papules, excoriation, and lichenification), severity of lesions (0-3), and pruritus. The scores range from 0 to 72 for the main symptoms of AD and from 0 to 18 for pruritus, giving a maximum possible score of 0 (no involvement) to 90 (maximum involvement), (0-0.9 clear, 1-8.9 mild, 9.0-29.9 moderate, 30.0-90 severe).

SECONDARY OUTCOMES:
evaluate the tacrolimus safety | 4 months
  assessment of treatment related toxicities; assessment of the incidence rate of burning
evaluation of tacrolimus safety | 4 months
  assessment of other tacrolimus related toxicity; the incidence rate of stinging sensation
evaluation of safety of tacrolimus | 4 months
  assessment of the degree of erythema using Eczema Area and Severity Index (EASI). The EASI is a composite score comprising ratings of the severity of erythema, oedema/induration/papulation, excoriations and lichenification; each on a scale from 0 to 3.
evaluate the hydrocortisone safety | 4 months
  assessment of the incidence rate of skin atrophy and skin infection.

CONTACTS AND LOCATIONS:
Overall Officials: Amal A. Mohamed, Principal Investigator — Department of Biochemistry, National Hepatology and Tropical Medicine Research institute
Locations (1):
- Dermatology Clinic of National Hepatology and Tropical Medicine Research Institute, Cairo, Egypt

REFERENCES:
- [Background] Alaiti S, Kang S, Fiedler VC, Ellis CN, Spurlin DV, Fader D, Ulyanov G, Gadgil SD, Tanase A, Lawrence I, Scotellaro P, Raye K, Bekersky I. Tacrolimus (FK506) ointment for atopic dermatitis: a phase I study in adults and children. J Am Acad Dermatol. 1998 Jan;38(1):69-76. doi: 10.1016/s0190-9622(98)70541-9. PMID 9448208
- [Background] Hanifin JM, Thurston M, Omoto M, Cherill R, Tofte SJ, Graeber M. The eczema area and severity index (EASI): assessment of reliability in atopic dermatitis. EASI Evaluator Group. Exp Dermatol. 2001 Feb;10(1):11-8. doi: 10.1034/j.1600-0625.2001.100102.x. PMID 11168575
- [Background] Reitamo S, Rustin M, Ruzicka T, Cambazard F, Kalimo K, Friedmann PS, Schoepf E, Lahfa M, Diepgen TL, Judodihardjo H, Wollenberg A, Berth-Jones J, Bieber T; European Tacrolimus Ointment Study Group. Efficacy and safety of tacrolimus ointment compared with that of hydrocortisone butyrate ointment in adult patients with atopic dermatitis. J Allergy Clin Immunol. 2002 Mar;109(3):547-55. doi: 10.1067/mai.2002.121832. PMID 11898005
- [Derived] Mohamed AA, El Borolossy R, Salah EM, Hussein MS, Muharram NM, Elsalawy N, Khalil MG, Mahmoud MO, El-Amir RY, Elsanhory HMA, Ahmed N, Adaroas AS, Montaser M, El Kholy AA. A comparative randomized clinical trial evaluating the efficacy and safety of tacrolimus versus hydrocortisone as a topical treatment of atopic dermatitis in children. Front Pharmacol. 2023 Sep 20;14:1202325. doi: 10.3389/fphar.2023.1202325. eCollection 2023. PMID 37799965